CLINICAL TRIAL: NCT06432686
Title: Neurophysiological Effects of Transcutaneous Electrical Nerve Stimulation in Persons With MS - a Pilot Study
Brief Title: Neurophysiological Effects of Transcutaneous Electrical Nerve Stimulation in Persons With MS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: MS-fMRI-TENS
Record Dates: First submitted 2024-05-22; First posted 2024-05-29 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Fatigue; Walking, Difficulty; Multiple Sclerosis
MeSH Terms: conditions — Fatigue; Mobility Limitation; Multiple Sclerosis | interventions — Transcutaneous Electric Nerve Stimulation; Movement

STUDY DESIGN:
Intervention Model Description: * sham stimulation of the tibialis anterior,
  * active stimulation of the tibialis anterior,
  * active stimulation of the quadriceps,
  * continuous movement of the foot (plantar & dorsiflexion),
  * a combination of sham stimulation of the tibialis anterior and movement of the foot,
  * a combination of stimulation of the tibialis anterior and movement of the foot.
  The order of these conditions is randomized.
Who Masked: Participant
Masking Description: All participants receive both active and sham TENS. Subjects will be told they will get two types of stimulation but they are not being told that one is 'sham' and the other 'active', to minimalize a placebo effect. Researchers are not blinded, but also interacting minimally with the participant while they are lying in the scanner.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (6):
- sham stimulation of the tibialis anterior (Sham Comparator)
  Interventions: Device: Transcutaneous Electrical Nerve Stimulation
- active stimulation of the tibialis anterior (Experimental)
  Interventions: Device: Transcutaneous Electrical Nerve Stimulation
- active stimulation of the quadriceps (Experimental)
  Interventions: Device: Transcutaneous Electrical Nerve Stimulation
- continuous movement of the foot (plantar & dorsiflexion) (Active Comparator)
  Interventions: Behavioral: Movement
- a combination of sham stimulation of the tibialis anterior and movement of the foot (Sham Comparator)
  Interventions: Device: Transcutaneous Electrical Nerve Stimulation; Behavioral: Movement
- a combination of active stimulation of the tibialis anterior and movement of the foot (Experimental)
  Interventions: Device: Transcutaneous Electrical Nerve Stimulation; Behavioral: Movement

INTERVENTIONS:
Device: Transcutaneous Electrical Nerve Stimulation — Transcutaneous electrical nerve stimulation (TENS) is a safe, relatively cheap, and non-painful stimulation of the peripheral sensory and motor nerves. The stimulator is easy to operate and pwMS can apply the stimulation themselves at home. This makes TENS an interesting tool to augment sensory input. A high frequency and long pulse duration is used.
  Arms: a combination of active stimulation of the tibialis anterior and movement of the foot; a combination of sham stimulation of the tibialis anterior and movement of the foot; active stimulation of the quadriceps; active stimulation of the tibialis anterior; sham stimulation of the tibialis anterior
Behavioral: Movement — Participants are instructed to perform plantar- and dorsi-flexion contraction in a relatively slow tempo. The movement of the ankle is measured by an MRI-compatible potentiometer and participants receive feedback of this movement on the screen inside the scanner.
  Arms: a combination of active stimulation of the tibialis anterior and movement of the foot; a combination of sham stimulation of the tibialis anterior and movement of the foot; continuous movement of the foot (plantar & dorsiflexion)

SUMMARY:
Transcutaneous Electrical Nerve Stimulation (TENS) is a treatment that could potentially reduce walking problems and fatigue in persons with Multiple Sclerosis. However, extensive use of TENS in a clinical setting is hindered by a lack of neurophysiological understanding of the effects of TENS. The primary objective of this pilot study is therefore to investigate the effects of TENS on brain activity in pwMS measured with fMRI.

DETAILED DESCRIPTION:
This study is an exploratory study to see if we can detect changes in fMRI activity during TENS in persons with MS. This is a randomized, single-blind crossover design. Subjects will undergo an MRI scan while they receive sham stimulation of the tibialis anterior, active stimulation of the tibialis anterior, stimulation of the quadriceps, perform continuous movements of the foot (plantar & dorsiflexion) and a combination of stimulation of the tibialis anterior and movement of the foot. This study will include 15 subjects with relapsing remitting or progressive MS and 15 healthy controls. Blood-oxygen-level-dependent (BOLD) activation changes and the interaction networks before, during and after active TENS and differences in activation due to stimulation on quadriceps vs. tibialis anterior, stimulation on tibialis anterior vs plantar/dorsiflexion and stimulation on tibialis anterior vs stimulation combined with plantar/dorsiflexion. This will be compared between pwMS and healthy controls. This study can add to the limited knowledge and possibly help to personalize and implement TENS in the clinic.

ELIGIBILITY:
Inclusion Criteria:

* age: 18-65 years
* EDSS score < 7

Exclusion Criteria:

* metal or electrical implants
* BMI > 40
* claustrophobia
* being pregnant
* having a psychiatric disorder
* having cognitive or communication problems which reduces the capacity to understand instructions
* having a neurological disorder other than MS
* having cardiac arrhythmia

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
BOLD activation due to TENS | 1 hour fMRI scan
  Blood level detection activation (BOLD) changes and interaction networks before, during and after active TENS and differences in activation due to stimulation on quadriceps vs. tibialis anterior, stimulation on tibialis anterior vs plantar/dorsiflexion and stimulation on tibialis anterior vs stimulation combined with plantar/dorsiflexion. We focus on the thalamus (integration station of sensory input), sensory cortex (sensory awareness) and motor cortices (sensorimotor integration).

IPD SHARING:
Plan to Share IPD: Undecided